CLINICAL TRIAL: NCT03492476
Title: Controlled, Randomized Clinical Trial of the Circaid® Compression Sleeve Versus Short-stretching Bandage at the Reduction Phase of Upper Limb Lymphatic Edema and Versus Compression Sleeve and Short-stretching Bandages at the Initial Maintenance Phase
Brief Title: Circaid® Compression Sleeve Versus Short-stretching Bandage in Upper Limb Lymphatic Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEN Biotech (Industry)
Collaborators: medi (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1512
Record Dates: First submitted 2018-03-22; First posted 2018-04-10 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Lymphedema of Upper Arm
Keywords: Lymphedema of Upper Arm reduction; Lymphedema Upper Arm device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circaid (Experimental): Compression sleeve on the day associated with the night wearing of the system of contention circaid®
  Interventions: Device: Circaid
- Reference treatment (Active Comparator): Compression sleeve during the day associated with a possible treatment with it during the night, according to the recommendations of the HAS
  Interventions: Device: Short-stretching Bandage (Reference treatment)

INTERVENTIONS:
Device: Circaid — Three observation periods were defined with the following products:
  * D1 to D5: intensive hospital treatment performed by the night and day wearing of the circaid® compression system
  * Day of Discharge (DD) from the hospital to DD +30: ambulatory initial maintenance phase carried out by the wearing of a compression sleeve on the day associated with the nighttime compression system circaid®
  * DD + 31 to DD + 90: ambulatory maintenance phase carried out by the wearing of a compression sleeve on the day associated with the nighttime circaid® compression system
  Other Names: Non-elastic bands
  Arms: Circaid
Device: Short-stretching Bandage (Reference treatment) — Three observation periods were defined with the following products:
  * D1 to D5: intensive hospital treatment performed by the night and day wearing of short stretching tapes.
  * DD (Day of discharge from the hospital) to DD +30: ambulatory initial maintenance phase carried out by the wearing of a compression sleeve on the day associated with a possible treatment at night, as recommended by HAS.
  * DD + 31 to DD + 90: ambulatory maintenance phase carried out by the wearing of a compression sleeve on the day associated with possible treatment at night
  Other Names: Non-elastic bands
  Arms: Reference treatment

SUMMARY:
One of the difficulties encountered in the treatment of lymphedema, both in the active reduction phase and in the maintenance phase, is the appliance of the short-length compression bandages which requires good technicality and experience to exert the pressure required to remove liquids from tissue spaces and reduce the volume of the arm or prevent it from increasing again.

The study aims to compare the current protocol of care considered optimal for the reduction of lymphedema and the maintenance of this reduction with the protocol of care which would integrate the device circaid® in substitution to the laying of bands with short extension as it is now in other countries.

DETAILED DESCRIPTION:
During the intensive decongestive treatment phase, which usually takes place in specialized lymphedema treatment departments, the staff are properly trained and have the required experience, but the appliance of these short-length compression bandages requires a lot of time. During the maintenance phase, the appliance of short stretch bandages gives way during the day to the wearing of a compression sleeve which can be put on fairly easily. But during the night, in the absence of a nurse or a spouse with the technical skills required to put them in place, few patients can benefit from the wearing of short stretching bandages. During the maintenance phase, many patients quickly give up these nocturnal bandages, thus losing the gain obtained during the reduction phase. This situation is all the more regrettable that, as shown in the studies, this nocturnal wearing contributes to a very significant reduction in the rate of reappearance of lymphedema and avoids the recurrent need of intensive reduction sessions in hospitals, which are costly for health insurance. and uncomfortable for the patients.

To improve this situation, medi has developed a device called circaid®, consisting of non-elastic bands adjustable and repositionable with "Velcro" systems, which can be used both for the intensive reduction phase but also during the maintenance phase by the patients themselves because of its ease of placement.

It is composed of several inelastic strips or removable straps, parallel and overlapping slightly to leave no crease and no space between them. Velcro tabs or fasteners help ensure proper initial positioning and readjustment as the arm volume is reduced. This gives a given pressure by tightening or loosening each band while limiting friction and discomfort. In the intensive reduction phase, its ease of use reduces the time devoted by nurses to the use of short stretching tapes which, in addition to the need for good technique, requires a significant amount of time. In the maintenance phase, this original and comfortable compression device allows the patient to become autonomous after minimal learning. The simplicity of the introduction of the system on the limb and the calibration of the delivered pressure allows to develop the self management of the treatment, because it is possible to reposition the bands as and when the decrease of the edema, which makes it possible to optimize the effectiveness of the treatment. The ability to instantly readjust the circaid®Juxtafit system allows to constantly apply the right level of pressure delivered, to reduce the volume of the limb. This is not possible with a traditional multilayer bandage if the different layers are not completely remove. A visual calibrator ensures the right level of pressure delivered at all times.

In addition to efficiency, patients' quality of life is improved by being able to remove and return it on their own, making it easier to wash or dress. Similarly, less rigid while being just as compressive, it allows a better comfort in the daily gestures and in particular to have a normal range of arm flexion movements more compatible with driving than the wearing of tapes.

The product is currently marketed in many countries and is reimbursed in the following countries: United States, Quebec, the Netherlands, United Kingdom, Austria in the indication of the treatment of lymphedema.

In view of its admission to reimbursement in France, a meeting was held with HAS experts in the context of the so-called early meeting procedure in order to define the study that should be done. A detailed synopsis which is the one of the present protocol has been validated by the methodological experts of the HAS as being able to bring the arguments of effectiveness required by being as close as possible to the usual practice and by covering at the same time the phase of intensive reduction and the maintenance phase. It aims to compare the current protocol of care considered optimal for the reduction of lymphedema and the maintenance of this reduction with the protocol of care which would integrate the device circaid® in substitution to the laying of bands with short extension as it is now in other countries.

ELIGIBILITY:
Inclusion Criteria:

* be women over the age of 18;
* presenting a unilateral lymphedema of the upper limb of stage II or III according to the International Society of Lymphology, secondary to the curative ganglion treatment of a cancer, whatever its nature, and requiring a decongestive treatment by contention / compression;
* presenting an increase in the volume of the arm affected by lymphedema of at least 10% when compared to the contralateral arm;
* benefiting of the French health insurance coverage;
* duly informed of the benefits, constraints and risks of the study;
* medically and legally able to understand the methods of carrying out the study and to give written informed consent to participate in the study;
* having given their free written informed consent to their participation in the study

Exclusion Criteria:

Not be included in the study:

* from a medical point of view, the patients:

  * with stage I lymphedema;
  * with lymphedema of multiple locations;
  * having had intensive decongestive treatment in the last 6 months;
  * having a recurrence of cancer or a peripheral arterial disease contraindicating or restraining compression.
* from a legal point of view, the patients:

  * not in a position to give free and informed consent because of an administrative or judicial decision or a pathology that may affect their judgment or a difficulty of linguistic comprehension;
  * currently participating in another clinical trial or in an exclusion period from another clinical trial;
  * who may not adhere to the terms of the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only can be recruited.
Enrollment: 142 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Volume reduction of upper limb lymphatic edema D30 | 30 days
  The main objective of the study is to compare, at the 30th day of the initial maintenance phase, the reduction in the volume of lymphatic edema of the upper limb obtained under the effect of the wearing of a compression sleeve on the day associated with the night wearing of the system of contention circaid® versus the wearing of a compression sleeve during the day associated with a possible treatment with it during the night, according to the recommendations of the french High Authority of Health (HAS).

SECONDARY OUTCOMES:
Volume reduction of upper limb lymphatic edema D5 | 5 days
  To compare, on the 5th day of the reduction phase, the reduction in the volume of lymphatic edema of the upper limb obtained under the effect of the night and day wearing of the circaid® compression system and the night and day wearing of short lengthening bands such as recommended by the HAS
Volume reduction of upper limb lymphatic edema D90 | 90 days
  To compare, at the 90th day of the maintenance phase, the reduction in the volume of lymphatic edema maintained by the wearing of a compression sleeve during the day associated with the circaid® compression system at night and the wearing of a compression sleeve during the day associated with a possible wearing at night.
Physician's opinion on lymphedema-induced discomfort improvement D5 (Clinical Global Improvement Impression) | 5 days
  To compare, at the 5th day of the reduction phase the physicians' opinions on lymphedema-induced discomfort improvement through the Clinical Global Improvement Impression (CGII). The evaluation focuses on the change in the volume of lymphoedema. The scale has 7 levels: from "Significantly decreased" (better outcome) to "Significantly increased" (worse outcome). Intermediate levels are: "Much decreased"; "Slightly decreased", "No change"; "Slightly increased"; "Much increased".
Patient's opinion on lymphedema-induced discomfort improvement D5 (Patient Global Improvement Impression) | 5 days
  To compare, at the 5th day of the reduction phase the patient's opinions on lymphedema-induced discomfort improvement through the Patient Global Improvement Impression (PGII). The evaluation focuses on the change in the volume of lymphoedema. The scale has 7 levels: from "Significantly decreased" (better outcome) to "Significantly increased" (worse outcome). Intermediate levels are: "Much decreased"; "Slightly decreased", "No change"; "Slightly increased"; "Much increased".
Patient's opinion on lymphedema-induced discomfort improvement D30 (Patient Global Improvement Impression) | 30 days
  To compare, at the 30th day of the reduction phase the patient's opinions on lymphedema-induced discomfort improvement through the PGII (Patient Global Improvement Impression). The evaluation focuses on the change in the volume of lymphoedema. The scale has 7 levels: from "Significantly decreased" (better outcome) to "Significantly increased" (worse outcome). Intermediate levels are: "Much decreased"; "Slightly decreased", "No change"; "Slightly increased"; "Much increased".
Patient's opinion on lymphedema-induced discomfort improvement D90 (Patient Global Improvement Impression) | 90 days
  To compare, at the 90th day of the reduction phase the patient's opinions on lymphedema-induced discomfort improvement through the PGII (Patient Global Improvement Impression). The evaluation focuses on the change in the volume of lymphoedema. The scale has 7 levels: from "Significantly decreased" (better outcome) to "Significantly increased" (worse outcome). Intermediate levels are: "Much decreased"; "Slightly decreased", "No change"; "Slightly increased"; "Much increased".
Physician's opinion on lymphedema-induced discomfort improvement D30 (Clinical Global Improvement Impression) | 30 days
  To compare, at the 30th day of the reduction phase the physicians' opinions on lymphedema-induced discomfort improvement through the CGII (Clinical Global Improvement Impression). The evaluation focuses on the change in the volume of lymphoedema. The scale has 7 levels: from "Significantly decreased" (better outcome) to "Significantly increased" (worse outcome). Intermediate levels are: "Much decreased"; "Slightly decreased", "No change"; "Slightly increased"; "Much increased".
Physician's opinion on lymphedema-induced discomfort improvement D90 (Clinical Global Improvement Impression) | 90 days
  To compare, at the 90th day of the reduction phase the physicians' opinions on lymphedema-induced discomfort improvement through the CGII (Clinical Global Improvement Impression). The evaluation focuses on the change in the volume of lymphoedema. The scale has 7 levels: from "Significantly decreased" (better outcome) to "Significantly increased" (worse outcome). Intermediate levels are: "Much decreased"; "Slightly decreased", "No change"; "Slightly increased"; "Much increased".
Patient's satisfaction about efficiency of the treatment D30 (Likert scale) | 30 days
  To compare, at the 30th day of the initial maintenance phase the patient's satisfaction. Patient assesses her satisfaction on a 5 items Likert scale from "Not at all efficient" (worse outcome) to "Very efficient" (better outcome). Intermediate levels are: "A bit"; "Moderately"; "Efficient".
Patient's satisfaction about wearing comfort of the treatment D30 (Likert scale) | 30 days
  To compare, at the 30th day of the initial maintenance phase the patient's wearing comfort experienced. Patient assesses her satisfaction on a 5 items Likert scale from "Not at all comfortable" (worse outcome) to "Very comfortable" (better outcome). Intermediate levels are:"A bit"; "Moderately"; "Comfortable".
Patient's satisfaction about efficiency of the treatment D90 (Likert scale) | 30 days
  To compare, at the 90th day of the initial maintenance phase the patient's satisfaction. Patient assesses her satisfaction on a 5 items Likert scale from "Not at all efficient" (worse outcome) to "Very efficient" (better outcome). Intermediate levels are: "A bit"; "Moderately"; "Efficient".
Patient's satisfaction about wearing comfort of the treatment D90 (Likert scale) | 90 days
  To compare, at the 90th day of the initial maintenance phase the patient's wearing comfort experienced. Patient assesses her satisfaction on a 5 items Likert scale from "Not at all comfortable" (worse outcome) to "Very comfortable" (better outcome). Intermediate levels are:"A bit"; "Moderately"; "Comfortable".
Patient's opinions on the ease of use of the product D90 (6 items to be completed by the patient) | 30 days
  To compare, at the 90th day of the initial maintenance phase the patients' opinions on the ease of use of the product. The patient have to complete 6 items (Yes/no response) : "Did you need caregiver's help ?"; "Did you need a third party to install the device ?"; "Did you have difficulty applying the required pressures ?"; "Do you wish to continue using the device ?"; "Would you recommend this device to third parties ?"; "Does the device seem easy to use ?".
Tolerance of the different products (patient evaluation on self-administered questionnaire) | 90 days
  To compare the tolerance of the different products at different phases of reduction and maintenance. Evaluation item on patient self-administered questionnaire "Intolerance to the device" to be assessed every week (Yes/no response, if yes, the patient have to precise).
Quality of patient's life assessment with the Lymphoedema Functioning, Disability and Health questionnaire (Lymph-ICF) | 90 days
  The quality of patient's life is assessed at each visit (D0, D5, D30, D90) with the Lymphoedema Functioning, Disability and Health questionnaire (Lymph-ICF).

CONTACTS AND LOCATIONS:
Overall Officials: MARLENE COUPE, MD, Study Chair — University Hospital, Montpellier; ERIC MARTIN, M., Study Director — medi France
Locations (4):
- France (4):
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Chu Saint Eloi, Montpellier
  - Ghr Mulhouse Sud Alsace, Mulhouse
  - Hopital Cognacq Jay, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paskett ED, Dean JA, Oliveri JM, Harrop JP. Cancer-related lymphedema risk factors, diagnosis, treatment, and impact: a review. J Clin Oncol. 2012 Oct 20;30(30):3726-33. doi: 10.1200/JCO.2012.41.8574. Epub 2012 Sep 24. PMID 23008299
- [Background] Leone N, Voirin N, Roche L, Binder-Foucard F, Woronoff AS, Delafosse P, Remontet L, Bossard N, Uhry Z. Projection de l'incidence et de la mortalité par cancer en France métropolitaine en 2015. Rapport technique. Saint-Maurice (Fra): Institut de veille sanitaire, 2015. 62 p
- [Background] Grosclaude P, Remontet L, Belot A, Danzon A, Rasamimanana C, Bossard N. Survie des personnes atteintes de cancer en France, 1989-2007 - Etude à partir des registres des cancers du réseau Francim. Saint-Maurice: Institut de veille sanitaire; 2013. 412 p
- [Background] Hayes SC, Janda M, Cornish B, Battistutta D, Newman B. Lymphedema after breast cancer: incidence, risk factors, and effect on upper body function. J Clin Oncol. 2008 Jul 20;26(21):3536-42. doi: 10.1200/JCO.2007.14.4899. PMID 18640935
- [Background] Campbell KL, Pusic AL, Zucker DS, McNeely ML, Binkley JM, Cheville AL, Harwood KJ. A prospective model of care for breast cancer rehabilitation: function. Cancer. 2012 Apr 15;118(8 Suppl):2300-11. doi: 10.1002/cncr.27464. PMID 22488704
- [Background] Velanovich V, Szymanski W. Quality of life of breast cancer patients with lymphedema. Am J Surg. 1999 Mar;177(3):184-7; discussion 188. doi: 10.1016/s0002-9610(99)00008-2. PMID 10219851
- [Background] Shih YC, Xu Y, Cormier JN, Giordano S, Ridner SH, Buchholz TA, Perkins GH, Elting LS. Incidence, treatment costs, and complications of lymphedema after breast cancer among women of working age: a 2-year follow-up study. J Clin Oncol. 2009 Apr 20;27(12):2007-14. doi: 10.1200/JCO.2008.18.3517. Epub 2009 Mar 16. PMID 19289624
- [Background] Framework L. Best practice for the management of lymphoedema: an international consensus. London: MEP Ltd; 2006
- [Background] Chang CJ, Cormier JN. Lymphedema interventions: exercise, surgery, and compression devices. Semin Oncol Nurs. 2013 Feb;29(1):28-40. doi: 10.1016/j.soncn.2012.11.005. PMID 23375064
- [Background] Quere I, Presles E, Coupe M, Vignes S, Vaillant L, Eveno D, Laporte S, Leizorovicz A; POLIT Study investigators. Prospective multicentre observational study of lymphedema therapy: POLIT study. J Mal Vasc. 2014 Jul;39(4):256-63. doi: 10.1016/j.jmv.2014.05.004. Epub 2014 Jun 12. PMID 24931830
- [Background] Lymphoedema Framework International consensus. Best Practice for the management of Lymphoedema London: MEP Ltd, 2006 and 2nd Edition 2012
- [Background] Vignes S, Porcher R, Arrault M, Dupuy A. Factors influencing breast cancer-related lymphedema volume after intensive decongestive physiotherapy. Support Care Cancer. 2011 Jul;19(7):935-40. doi: 10.1007/s00520-010-0906-x. Epub 2010 May 22. PMID 20495983

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT03492476/Prot_SAP_000.pdf